CLINICAL TRIAL: NCT05131360
Title: Reducing Daily Stress Among Sexual and Gender Minorities (the REDUCE Study)
Brief Title: Reducing Daily Stress Among Sexual and Gender Minorities
Acronym: REDUCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-FY2020-4338
Record Dates: First submitted 2021-10-05; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-07

CONDITIONS: Social Discrimination; Sexual and Gender Minorities; Mindfulness
Keywords: Social stress; Stress from discrimination; Mindfulness; Anxiety; Depression; Sexual and gender minorities
MeSH Terms: conditions — Social Discrimination; Coitus; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Introduction Only (Placebo Comparator): This is the control; participants only partake in one day's worth of the introduction or foundational mindfulness activities on the HMI app.
  Interventions: Behavioral: Introduction Only
- Purpose Only (Experimental): Participants partake in the introduction or foundational mindfulness for one day and then perform purpose-based mindfulness techniques for 5 days on the HMI app.
  Interventions: Behavioral: Purpose Only
- Connection Only (Experimental): Participants partake in the introduction or foundational mindfulness for one day and then perform connection-based mindfulness techniques for 5 days on the HMI app.
  Interventions: Behavioral: Connection Only
- Connection and Purpose (Experimental): Participants partake in the introduction or foundational mindfulness for one day and then perform connection and purpose-based mindfulness techniques for 5 days on the HMI app.
  Interventions: Behavioral: Connection and Purpose
- Awareness Only (Experimental): Participants partake in the introduction or foundational mindfulness for one day and then perform awareness-based mindfulness techniques for 5 days on the HMI app.
  Interventions: Behavioral: Awareness Only
- Awareness and Purpose (Experimental): Participants partake in the introduction or foundational mindfulness for one day and then perform awareness and connection-based mindfulness techniques for 5 days on the HMI app.
  Interventions: Behavioral: Awareness and Purpose
- Awareness, Purpose, and Connection (Experimental): Participants partake in the introduction or foundational mindfulness for one day and then perform connection, awareness, and purpose-based mindfulness techniques for 5 days on the HMI app.
  Interventions: Behavioral: Awareness, Purpose, and Connection
- Awareness and Connection (Experimental): Participants partake in the introduction or foundational mindfulness for one day and then perform awareness and connection-based mindfulness techniques for 5 days on the HMI app.
  Interventions: Behavioral: Awareness and Connection

INTERVENTIONS:
Behavioral: Introduction Only — This is the placebo condition in which participants engage in one day of introductory mindfulness activities.
  Arms: Introduction Only
Behavioral: Purpose Only — Participants engage in one day of introductory mindfulness activities followed up by 5 days of purpose-based mindfulness techniques.
  Arms: Purpose Only
Behavioral: Connection Only — Participants engage in one day of introductory mindfulness activities followed up by 5 days of connection-based mindfulness techniques.
  Arms: Connection Only
Behavioral: Connection and Purpose — Participants engage in one day of introductory mindfulness activities followed up by 5 days of connection and purpose-based mindfulness techniques.
  Arms: Connection and Purpose
Behavioral: Awareness Only — Participants engage in one day of introductory mindfulness activities followed up by 5 days of awareness-based mindfulness techniques.
  Arms: Awareness Only
Behavioral: Awareness and Purpose — Participants engage in one day of introductory mindfulness activities followed up by 5 days of awareness and purpose-based mindfulness techniques.
  Arms: Awareness and Purpose
Behavioral: Awareness, Purpose, and Connection — Participants engage in one day of introductory mindfulness activities followed up by 5 days of awareness, connection, and purpose-based mindfulness techniques
  Arms: Awareness, Purpose, and Connection
Behavioral: Awareness and Connection — Participants engage in one day of introductory mindfulness activities followed up by 5 days of awareness and connection-based mindfulness techniques.
  Arms: Awareness and Connection

SUMMARY:
The purpose of this study is to identify which mindfulness technique, or combination of mindfulness techniques, is most effective at mediating or eliminating stress in emerging adults who are sexual and gender as well as racial or ethnic minorities. Participants will be randomly assigned to one of eight conditions that are composed of the mindfulness techniques of Awareness, Purpose, and Connection.

DETAILED DESCRIPTION:
Underrepresented racial/ethnic sexual and gender minorities (SGM) aged 18-29 will be recruited via convenience sampling from social media websites (e.g. Facebook, Instagram) and listservs from NYU student groups and through LGBT community partners. Interested persons who screen eligible through the study's online eligibility screener will be asked to provide their phone number and/or email address to be contacted by a research assistant. An online meeting via Zoom will then be scheduled to confirm eligibility, provide additional information concerning study parameters. The online meeting will be between the research assistant and a single participant. The meeting will take between 10 to 15 minutes depending on the questions individuals may have. The meeting will be an informational assessment to assure that the individual can effectively use and have access to the materials used in the study, the online surveys/assessments, and interventions.

After providing online informed consent through REDCap, the participant will be randomized into one of the 8 mindfulness conditions, complete a 30-minute baseline survey via REDCap, and be provided with training on study protocols. Participants will engage in the study of a 5-day period (starting after the baseline survey). Participants will engage in one of 8 interventions, depending on randomization, in which participants will engage with mindfulness activities each night for a total of 5 nights which is expected to take 10-20 minutes per day (the exception to this is the control condition who only receives an introduction to mindfulness on day 1). In addition, each night over the 5-day period, participants will be sent a REDCap survey to complete a "nightly diary" which will take about 5 minutes to complete.

After completion of the 5-day protocol, participants will be scheduled for an online Zoom meeting where participants will engage in a 30-40 minute debrief interview and be renumerated. The Zoom meetings will be between a research assistant and a single participant. Lastly, in order to improve retention, RA's will perform check-in calls twice during the 5-day daily diary period.

The interventions will be administered using the multiphase optimization strategy (MOST). The participants will be randomized to at least one of the 3 intervention components of Awareness, Purpose, and Connection for this optimization study, which make up the 8 conditions. Each of these components is known to be effective in reducing stress and promoting well-being among populations that experience a high rate of discrimination (e.g., SGM). The three components are administered via the Healthy Minds Program (HMP), which is a smartphone app-based mindfulness intervention developed through the research of Dr. Richard Davidson and his team at the University of Wisconsin-Madison's Center for Healthy Minds in affiliation with the non-profit Healthy Minds Innovations (HMI). The app provides an average of 10-minute meditations that can be completed while sitting, walking, or exercising that focus on the modules of Awareness, Purpose, and Connection. Participants will log into the app and listen to the meditations that correspond to their selected randomization on each of the 5 days. The app's methodology aligns with constituents of psychological well-being that are trainable and measurable as evidenced by the Center for Healthy Minds: Awareness, Purpose, and Connection. The components are as follows: 1) Awareness through meditation promotes self-awareness, reducing the mind's ability to be distracted and instead be present at the moment. Awareness promotes well-being by bringing attention to the present moment, not allowing the mind to wander to negative thoughts that cause stress; 2) Purpose through meditation promotes mindfulness of one's thoughts and feelings in the present moment and encourages compassion with oneself and positive reappraisal; 3) Connection through meditation supports empathy, compassion, and kindness in daily activities. By shifting to this positive mindset, individuals are able to cultivate social support networks which research has found to decrease the risk for depression.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-29 years
* Must identify as a sexual minority (e.g. gay, bisexual, sexually fluid, etc.)
* Must identify as an underrepresented racial/ethnic minority
* Have an active cell phone service and be able to access the cell phone 7 days a week between 6 p.m. and 6 a.m. the next morning
* Be willing and able to receive up to 6 text messages per day
* Have consistent Internet access 7 days a week between 6 p.m. and 6 a.m.
* Can understand, read, and speak English
* Willing to provide written informed consent.

Exclusion Criteria:

* Not between 18-29 years
* Does not identify as a sexual minority (e.g. gay, bisexual, sexually fluid, etc.)
* Does not identify as an underrepresented racial/ethnic minority
* Does not have an active cell phone service and or ability to access the cell phone 7 days a week between 6 p.m. and 6 a.m. the next morning
* Not willing and able to receive up to 6 text messages per day
* Does not have consistent Internet access 7 days a week between 6 p.m. and 6 a.m.
* Does not have the ability to understand, read, and speak English
* Not willing to provide written informed consent.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Perceived Stress on the Perceived Stress Scale at Day 5 | Baseline through study completion, up to one year
  The primary outcome for this study is change in perceived stress as measured by the Perceived Stress Scale from baseline to Day 5 among all study participants.
Change from Baseline in Satisfaction with Life on the Satisfaction with Life Scale at Day 5 | Baseline through study completion, up to one year
  The primary outcome for this study is change in perceived satisfaction with life as measured by the Satisfaction with Life Scale from baseline to Day 5 among all study participants.

SECONDARY OUTCOMES:
Optimized Intervention Package | Through study completion, an average of 1 year
  An optimal intervention combination will be determined with the primary outcomes of perceived stress (as measured through the Perceived Stress Scale) and satisfaction with life (as measured through the Satisfaction with Life Scale) by looking at changes in mean perceived stress and satisfaction with life across all intervention categories.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie H Cook, DrPH, Principal Investigator — New York University
Locations (1):
- New York University School of Global Public Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
N/A (not to be shared with other researchers)

REFERENCES:
- [Derived] Cook SH, Wood EP, Mirin N, Bandel M, Delorme M, Gad L, Jayakar O, Mustafa Z, Tatar R, Javdani S, Godfrey E. A Mindfulness-Based Intervention to Alleviate Stress From Discrimination Among Young Sexual and Gender Minorities of Color: Protocol for a Pilot Optimization Trial. JMIR Res Protoc. 2022 Jan 14;11(1):e35593. doi: 10.2196/35593. PMID 34928237

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT05131360/Prot_SAP_ICF_000.pdf